CLINICAL TRIAL: NCT02598089
Title: A Phase 1 Double Blinded, Randomized, Placebo-Controlled Study In Healthy Adult Volunteers In Vietnam To Examine The Safety And Immunogenicity Of A Seasonal Trivalent Inactivated Split Virion Influenza Vaccine (IVACFLU-S) Produced By IVAC
Brief Title: Seasonal Trivalent Inactivated Split Virion Influenza Vaccine Clinical Trial (IVACFLU-S)
Acronym: IVACFLU-S
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Vaccines and Medical Biologicals, Vietnam (Industry)
Collaborators: National Institute of Hygiene and Epidemiology, Vietnam (Other); World Health Organization (Other); Department of Health and Human Services (U.S. Federal Agency); PATH (Other); Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IVACFLU-S-01; NCT02809209 (obsolete NCT alias)
Record Dates: First submitted 2015-10-15; First posted 2015-11-05 (Estimated); Results first posted 2019-01-28 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Influenza, Human
Keywords: Seasonal Influenza; Trivalent Vaccine; Inactivated Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trivalent Seasonal Influenza Vaccine (Experimental): 0.5 mL of seasonal trivalent influenza vaccine with 15 mcg of HA of each of 3 strains:
  * NYMC BX-51B reassortant of B/Massachusetts/2/2012
  * NYMC X-179A reassortant of A/California/7/2009 (H1N1)
  * NYMC X-223A reassortant of H3/A/Texas/50/2012 (H3N2)
  Interventions: Biological: Trivalent Seasonal Influenza Vaccine
- Placebo (Placebo Comparator): This is the placebo comparator: 0.5 mL of Phosphate Buffered Saline
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Trivalent Seasonal Influenza Vaccine
  Other Names: IVACFLU-S
  Arms: Trivalent Seasonal Influenza Vaccine
Other: Placebo — 0.5 mL of phosphate buffered saline
  Arms: Placebo

SUMMARY:
This is a phase I, double-blind, randomized, placebo-controlled trial with two groups of subjects to receive seasonal trivalent inactivated split virion influenza vaccine (A/H1N1; A/H3N2 and B strains) or placebo (phosphate buffered saline). A total of 60 healthy male and female adults 18 through 45 years of age will be randomized to receive vaccine (30) or placebo (30).

DETAILED DESCRIPTION:
This is a phase 1, single center, double blinded, randomized, placebo-controlled study. Sixty (60) healthy male and female adults, 18 to 45 years of age, will be enrolled into the trial. Subjects will be randomized 1:1 to one of two treatment allocations: 30 to vaccine, 30 to placebo. The study will utilize a "randomized block design" to assure a balance of 1:1 vaccine and placebo when all subjects are enrolled. The study will be double blinded, meaning the study subjects, investigators, and the sponsor will be unaware of the treatment allocated to each subject until the clinical trial database is declared final and locked. The study should take about 5 months to complete, with each subject involved for 3 months from the day of injection. The justification for the 3 month follow up, rather than 6 month follow up is that this is an inactivated vaccine that follows very standard manufacturing practices with standard antigens. The safety of inactivated influenza vaccines is well-established. Adding length to the follow up results in delays in future testing of the vaccine for licensure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult 18 through 45 years of age at the enrollment visit.
* Literate (by self-report) and willing to provide written informed consent.
* Healthy, as established by the medical history, physical examination, and screening laboratory evaluations.
* Capable and willing to complete Diary Cards and willing to return for all follow-up visits.
* For females, willing to utilize reliable birth control measures (e.g., intrauterine device, hormonal contraception, condoms) through the Day 22 visit.

Exclusion Criteria:

* Participation in another clinical trial involving any therapy within the previous three months or planned enrollment in such a trial during the period of this study.
* Receipt of any non-study vaccine within 4 weeks prior to enrollment or refusal to postpone receipt of such vaccines until after the Day 22 visit.
* Current or recent (within 2 weeks of enrollment) acute illness with or without fever.
* Receipt of immune globulin or other blood products within 3 months prior to study enrollment or planned receipt of such products prior to the Day 22 visit.
* Chronic administration (defined as more than 14 consecutively-prescribed days) of immunosuppressants or other immune-modulating therapy within six months prior to study enrollment. (For corticosteroids, this means prednisone or equivalent, 0.5 mg per kg per day; topical steroids are allowed.)
* History of asthma.
* Hypersensitivity after previous administration of any vaccine.
* Suspected or known hypersensitivity to any of the study vaccine components, including chicken or egg protein, antibiotics, and rubber (from the vaccine vial stoppers).
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatobiliary, metabolic, neurologic, psychiatric or renal functional abnormality, as determined by medical history, physical examination or clinical laboratory screening tests, which in the opinion of the investigator, might interfere with the study objectives.
* History of any blood or solid organ cancer.
* History of thrombocytopenic purpura or known bleeding disorder.
* History of seizures.
* Known or suspected immunosuppressed or immunodeficient condition of any kind.
* Confirmed hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Known human immunodeficiency virus (HIV) infection (self-report).
* Known active tuberculosis or symptoms of active tuberculosis, regardless of cause (self-report).
* History of chronic alcohol abuse and/or illegal drug use.
* Pregnancy or lactation. (A negative pregnancy test will be required before administration of study product for all women of childbearing potential.)
* History of Guillain-Barré Syndrome
* Any condition that, in the opinion of the investigator, would increase the health risk to the subject if he/she participates in the study or would interfere with the evaluation of the study objectives.

Note: Minor out-of-range laboratory values no greater than Grade 1 will not be considered to be exclusionary at screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dang D. Anh, Ph. D, Principal Investigator — National Institute of Hygiene and Epidemiology, Vietnam
Locations (1):
- Hung Ha District Health Center, Thái Bình, Thai Binh Province, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Anh DD, Thiem VD, Anh NTH, Huong VM, Nga NT, Thang TC, Thai DH, Chien VC, Holt R, Wahid R, Flores J, Berlanda Scorza F, Taylor DN. Randomized safety and immunogenicity trial of a seasonal trivalent inactivated split virion influenza vaccine (IVACFLU-S) in healthy young Vietnamese adults. Vaccine. 2016 Oct 26;34(45):5457-5462. doi: 10.1016/j.vaccine.2016.08.052. Epub 2016 Aug 24. PMID 27567493
- See also: Article published in the journal Vaccine — https://www.ncbi.nlm.nih.gov/pubmed/27567493

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixty four (64) subjects were consented and 4 were not randomized, leaving 60 subjects for the study.
Groups:
- Trivalent Seasonal Influenza Vaccine: 0.5 mL of seasonal trivalent influenza vaccine with 15 mcg of HA of each of 3 strains: B, H1N1 & H3N2
Period: Overall Study
Arm/Group | Trivalent Seasonal Influenza Vaccine | Placebo
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Trivalent Seasonal Influenza Vaccine: 0.5 mL of seasonal trivalent influenza vaccine with 15 mcg of HA of each of 3 strains: B, H1N1, & H3N2
- Total: Total of all reporting groups
Arm/Group | Trivalent Seasonal Influenza Vaccine | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Full Range); unit: years] | 37.7 [27 to 45] | 37.8 [21 to 45] | 37.8 [21 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 21 | 48
  Male | 3 | 9 | 12
Race/Ethnicity, Customized [Number; unit: participants]
  Kinh | 30 | 30 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 30 | 30 | 60
  Other | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Vietnam | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Immediate Adverse Events
Description: Any adverse event occurring within the 30 minute post vaccination period.
Time Frame: 30-minute post-vaccination period.
Population: The analysis was conducted for subjects who were randomized and received a study vaccination.
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Vaccine Group: 0.5 mL of influenza vaccine split, inactivated with 15 mcg of HA of each of 3 strains: B, H1N1, & H3N2
- Placebo Group: 0.5 mL of phosphate buffered saline
Arm/Group | Vaccine Group | Placebo Group
Number analyzed (Participants) | 30 | 30
participants | 0 [0 to 0] | 0 [0 to 0]

2. Primary Outcome: Number and Percentage of Participants Reporting Solicited Local Reactogenicity
Description: Number of subjects reporting solicited local reactions (redness, swelling, pain, hardness, and tenderness) at the injection site post-vaccination with study vaccine or placebo.
Time Frame: 7-day period (Days 1-7) post-vaccination.
Population: The analysis was conducted for subjects who were randomized and received a study vaccination
Measure: Count of Participants; unit: Participants
Groups:
- Vaccine Group: 0.5 mL of seasonal trivalent influenza vaccine with 15 mcg of HA of each of 3 strains: B, H1N1, & H3N2
Arm/Group | Vaccine Group | Placebo Group
Number analyzed (Participants) | 30 | 30
Participants
  Pain: Mild | 17 | 5
  Pain: Moderate | 2 | 0
  Pain: Severe | 0 | 0
  Pain: None | 11 | 25
  Tenderness: Mild | 16 | 9
  Tenderness: Moderate | 1 | 0
  Tenderness: Severe | 0 | 0
  Tenderness: None | 13 | 21
  Hardness: Mild | 0 | 0
  Hardness: Moderate | 1 | 0
  Hardness: Severe | 0 | 0
  Hardness: None | 29 | 30
  Swelling: Mild | 0 | 0
  Swelling: Moderate | 1 | 0
  Swelling: Severe | 0 | 0
  Swelling: None | 29 | 30
  Redness: Mild | 0 | 0
  Redness: Moderate | 0 | 0
  Redness: Severe | 0 | 0
  Redness: None | 30 | 30

3. Primary Outcome: Number and Percentage of Participants Reporting Solicited Systemic Reactogenicity
Description: Number of subjects reporting solicted systemic reactions (fever, fatigue/malaise, muscle aches, joint aches, chills, nausea, vomiting, and headache) post-vaccination with study vaccine or placebo
Time Frame: 7-day period (Days 1-7) post-vaccination
Population: The analysis was conducted for subjects who were randomized and received a study vaccination
Measure: Count of Participants; unit: Participants
Groups:
- Vaccine Group: 0.5 mL of seasonal trivalent influenza vaccine with 15 mcg of each of 3 strains: B, H1N1, & H3N2
Arm/Group | Vaccine Group | Placebo Group
Number analyzed (Participants) | 30 | 30
Participants
  Headache: Mild | 6 | 8
  Headache: Moderate | 1 | 1
  Headache: Severe | 0 | 0
  Headache: None | 23 | 21
  Tiredness/discomfort: Mild | 5 | 6
  Tiredness/discomfort: Moderate | 2 | 1
  Tiredness/discomfort: Severe | 0 | 1
  Tiredness/discomfort: None | 23 | 22
  Chills: Mild | 2 | 3
  Chills: Moderate | 0 | 1
  Chills: Severe | 0 | 0
  Chills: None | 28 | 26
  Muscle aches: Mild | 3 | 4
  Muscle aches: Moderate | 0 | 1
  Muscle aches: Severe | 0 | 0
  Muscle aches: None | 27 | 25
  Vomiting: Mild | 1 | 1
  Vomiting: Moderate | 0 | 0
  Vomiting: Severe | 0 | 0
  Vomiting: None | 29 | 29
  Joint aches: Mild | 0 | 1
  Joint aches: Moderate | 1 | 0
  Joint aches: Severe | 0 | 1
  Joint aches: None | 29 | 28
  Nausea: Mild | 0 | 3
  Nausea: Moderate | 0 | 0
  Nausea: Severe | 0 | 0
  Nausea: None | 30 | 27

4. Primary Outcome: Number and Percentage of Participants With Unsolicited Adverse Events
Description: Unsolicited AEs were any AEs that occurred any time after the vaccine/placebo was administered (temporally related to investigational product), whether or not deemed "related" to the product, and are not solicited (specifically asked of the subject). Unsolicited AEs were to be observed by the study center personnel while the subject was at the study center for a study visit or reported by the subject at any time. Any sign or symptom that would normally be considered a "solicited AE" (for example, fever, nausea, injection site pain) starting after 7 days post-vaccination were to be recorded as an "unsolicited AE. In this study, laboratory results were considered AEs when (1) the result was judged to be clinically significant by the Principal Investigator, regardless of grade; or (2) the result is Grade 2 or higher.
  Note: all unsolicited AEs were mild in intensity. Please see Adverse Events section of this report for detailed information of AEs.
Time Frame: Within 21 days post-vaccination
Population: The analysis was conducted for subjects who were randomized and received a study vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- Vaccine Group: 0.5 mL of seasonal influenza vaccine with 15 mcg of HA of each of 3 strains: B, H1N1, & H3N2
Arm/Group | Vaccine Group | Placebo Group
Number analyzed (Participants) | 30 | 30
Participants | 7 | 7

5. Primary Outcome: Number and Percentage of Participants With Serious Adverse Events (SAEs)
Time Frame: Over the entire study period (Day 91)
Population: The analysis was conducted for subjects who were randomized and received a study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Group | Placebo Group
Number analyzed (Participants) | 30 | 30
Participants
  Serious Adverse Events (SAEs)--related | 0 | 0
  SAEs--not related | 0 | 0

6. Secondary Outcome: Number and Percentage of Subjects With Seroconversion Against Each of the 3 Antigens
Description: Seroconversion is defined as a serum HAI titer meeting the following criteria:
  * pre-vaccination titer <1:10 and a post-vaccination titer ≥ 1:40 or
  * pre-vaccination titer ≥ 1:10 and at least a four-fold increase in post-vaccination measured on Day 22.
Time Frame: Day 22
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Group | Placebo Group
Number analyzed (Participants) | 30 | 30
Participants
  Seroconversion rate to H1N1 | 28 | 0
  Seroconversion rate to H3N2 | 25 | 0
  Seroconversion rate to B | 23 | 0

7. Secondary Outcome: Number and Percentage of Seroprotected Subjects Against 3 Strains of Influenza Vaccine
Description: A seroprotected subject was defined as a vaccinated subject who had a serum Hemagluttination Inhibition (HAI) titer >/= 1:40. The 3 influenza strains assessed were B, H1, and H3.
Time Frame: Day 1 and Day 22 post vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Group | Placebo Group
Number analyzed (Participants) | 30 | 30
Participants
  H1 | 29 | 6
  H3 | 29 | 16
  B | 28 | 0

8. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Hemaggluntination Inhibition (HAI) Antibodies for Each Antigen
Description: Geometric mean titers (GMTs) of Serum Hemaggluntination Inhibition (HAI) antibodies pre- (Day 1) and post-vaccination (Day 22) for each of the 3 antigens.
Time Frame: Pre- (Day 1) and post-vaccination (Day 22)
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Placebo: 0.5 mL of Phosphate Buffered Saline
  Placebo Comparator: Placebo (PBS)
Arm/Group | Trivalent Seasonal Influenza Vaccine | Placebo
Number analyzed (Participants) | 30 | 30
Titers
  GMT to H1 Day 1 | 10.0 [6.7 to 15.0] | 10.6 [7.1 to 15.7]
  GMT to H1 Day 22 | 371.9 [245.4 to 563.6] | 10.7 [7.2 to 15.9]
  GMT to H3 Day 1 | 39.5 [22.9 to 68.4] | 35.6 [21.8 to 58.3]
  GMT to H3 Day 22 | 640 [419.2 to 977.1] | 33.6 [21.6 to 52.4]
  GMT to B Day 1 | 8.8 [6.7 to 11.6] | 6.9 [5.8 to 8.2]
  GMT to B Day 22 | 68.1 [47.1 to 98.2] | 7.0 [5.9 to 8.3]

9. Secondary Outcome: Geometric Mean Fold Rises (GMFRs) of Serum Hemaggluntination Inhibition (HAI) Antibodies
Description: Geometric mean fold rises (GMFRs) of serum hemaggluntination inhibition (HAI) antibodies post-vaccination/pre-vaccination for each of the 3 antigens
Time Frame: Day 22/Day1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Trivalent Seasonal Influenza Vaccine | Placebo
Number analyzed (Participants) | 30 | 30
fold rise
  GMFR Day 22/Day 1 for H1 | 37.2 [23.7 to 58.3] | 1 [0.9 to 1.0]
  GMFR Day 22/Day 1 for H3 | 16.2 [9.2 to 28.4] | 1.0 [0.9 to 1.0]
  GMFR Day 22/Day 1 for B | 7.7 [5.0 to 12.1] | 1.0 [0.9 to 1.0]

10. Secondary Outcome: Geometric Mean Neutralization Titers of Neutralizing Antibodies (MNT) Pre- (Day 1) and Post-Vaccination (Day 22) for Each of the 3 Antigens
Time Frame: Pre- (Day 1) and Post-vaccination (Day 22)
Population: All vaccinated subjects who have valid post vaccination immunogenicity measures with no major protocol deviations
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Vaccine Group | Placebo Group
Number analyzed (Participants) | 30 | 30
Titers
  GMT to H1 Day 1 | 8.7 [6.0 to 12.5] | 10.8 [7.3 to 16.1]
  GMT to H1 Day 22 | 417.4 [263.0 to 662.4] | 10.5 [7.2 to 15.3]
  GMT to H3 Day 1 | 38.6 [22.4 to 63.8] | 40.0 [23.5 to 68.1]
  GMT to H3 Day 22 | 670.3 [405.9 to 1106.7] | 39.1 [23.1 to 66.2]
  GMT to B Day 1 | 16.2 [10.3 to 25.6] | 14.6 [10.4 to 20.6]
  GMT to B Day 22 | 201.6 [123.6 to 328.8] | 14.3 [10.2 to 20.0]

11. Secondary Outcome: Geometric Fold Rises (GMFRs) of Neutralizing Antibodies (MNT) Post-vaccination/Pre-vaccination for Each of the 3 Antigens
Time Frame: Pre- (Day 1) and Post-vaccination (Day 22)
Population: All vaccinated subjects who have valid post-vaccination immunogenicity measures with no major protocol violations
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Vaccine Group | Placebo Group
Number analyzed (Participants) | 30 | 30
fold rise
  GMFR for H1 | 47.9 [29.1 to 79.0] | 1.0 [0.9 to 1.0]
  GMFR for B | 12.4 [6.9 to 22.3] | 1.0 [0.9 to 1.0]
  GMFR for H3 | 17.3 [9.7 to 31.0] | 1.0 [0.9 to 1.0]

ADVERSE EVENTS:
Time Frame: 90 days
Description: We included AEs that occurred any time after the vaccine/placebo was administered , whether or not deemed "related" to the product, and are not solicited (specifically asked of the subject) unless they started after 7 days post-vaccination. In this study, laboratory results were considered AEs when (1) the result was judged to be clinically significant by the Principal Investigator, regardless of grade; or (2) the result is Grade 2 or higher.
  Note: all unsolicited AEs were mild in intensity.
Arm/Group | Trivalent Seasonal Influenza Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 2/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trivalent Seasonal Influenza Vaccine (N=30) | Placebo (N=30)
Oropharyngeal pain/sore throat (Infections and infestations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No